CLINICAL TRIAL: NCT03674086
Title: Evaluation of the eAdjust Application to Provide Benefits in Users of Smartphone-connected Hearing Aids
Brief Title: Evaluation of the eAdjust Application
Status: Completed | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: Sonova AG (Industry); University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 18IH002
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2019-03

CONDITIONS: Hearing Loss, Bilateral; Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Bilateral; Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First-time hearing aid user: Using hearing aids less than or equal to three months.
  Interventions: Device: eAdjust 0.2 hearing aid smartphone application (or app)
- Existing hearing aid user: Using hearing aids for 6 months or more.
  Interventions: Device: eAdjust 0.2 hearing aid smartphone application (or app)

INTERVENTIONS:
Device: eAdjust 0.2 hearing aid smartphone application (or app) — The app connects to the Audeo B-90 Direct hearing aids via Bluetooth. The intended use for the app to enable hearing aid users to fine-tune their hearing aids. The app contains a series of sound modifiers, factory presets, sound modifier presets.

SUMMARY:
Despite being effective, the majority of people who would benefit from using hearing aids do not access them. For those who do obtain hearing aids, around 20% do not wear them regularly. People often do not use their hearing aids because they continue to experience difficulties when listening to and understanding speech in noisy situations.

Conventional hearing aids must be programmed and adjusted by a trained audiologist with specialist equipment and therefore provide limited user-control over the hearing aid's functionality. In comparison to conventional hearing aids, Smartphone-connected hearing aids enable patients to adjust their programmes themselves in different situations using a Smartphone application. Smartphone-connectivity can supplement clinical practices, as patients can adjust their hearing aids without the need to visit the clinic. This has the potential to empower patients to be actively involved in their own hearing healthcare.

A systematic review assessing the effectiveness of alternative listening devices showed that there is no published high-quality research assessing the clinical effectiveness of Smartphone-connected hearing aids. Furthermore, a usability research study has shown that patients want to personalise and adjust their own HA programmes to meet their individual needs. Having carried out the early development work, the next step would be to carry out a study to evaluate smartphone-connected hearing aids, in accordance with the MRC guidelines on developing and evaluating complex interventions.

This study will assess the benefits of a smartphone application, eAdjust that has been developed for use with Phonak Audeo B90-Direct hearing aids. The eAdjust app connects to the hearing aid via Bluetooth, and enables hearing aid users to fine-tune their hearing aids via their smartphone. The benefits of the eAdjust app will be assessed in the real-world as well as in the laboratory. A mixed methods approach will be taken, using both behavioural and patient reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years.
* With hearing loss type: symmetric (not more than 20 dB difference) and sensorineural.
* With mild to severe hearing loss in the categories: N2, N3, N4, N5, S2 and S3.
* No disturbing tinnitus.
* No contraindications against wearing hearing aids (e.g. ear disease or motor impairment).
* Hearing aid user:

  1. First-time (using hearing aids < 3 months)
  2. Existing (using hearing aids > 6 months)
* Owns an iPhone (v5 and IOS 10 or higher) and uses functions of her/his smartphone which exceed calling and writing text messages.
* Willing to wear test hearing aids, to use the eAdjust App, to take notes about experiences and to perform various tasks during the study period.
* English as a first spoken language or a good understanding of English. It is important that participants can understand the content of the resources and work with the interactive elements, as well as be able to answer outcome questionnaires, to ensure valid data are collected.

Exclusion Criteria:

- Unable to complete the questionnaires without assistance due to age-related problems (e.g. cognitive decline or dementia), to ensure valid data are collected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hearing aid users (first-time and existing) will be recruited from Nottingham Audiology Adult Service, Nottingham University Hospitals NHS Trust (secondary care). Immediately following the patient's hearing assessment appointment, a member of the patient's usual care team (audiologist) will identify eligible patients.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Hearing Handicap Inventory for the Elderly | Change from Baseline following 7-weeks of intervention use.
  25-item self-reported questionnaire assessing the effects of hearing loss on the emotional and social/situational adjustment. Scored using a three-point scale.

SECONDARY OUTCOMES:
Glasgow Hearing Aid Benefit Profile | Baseline (Part I) and following 7-weeks of intervention use (Part II).
  Assesses self-reported hearing disability and handicap (Part I), as well as hearing aid use, benefit, residual disability and satisfaction (Part II). Each domain is measured on a five-point scale.
Vanderbilt Fatigue Scale for Adults with Hearing Loss | Change from Baseline following 7-weeks of intervention use.
  A 40-item self-report measure of listening effort and fatigue. Scored using a five-point scale.
Device-Orientated Subjective Outcome scale | Change from Baseline following 7-weeks of intervention use.
  Self-report questionnaire suitable for quantifying subjective hearing aid outcomes. Scored using a seven-point response scale.
Glasgow Hearing Aid Difference Profile (existing hearing aid users only) | Change from Baseline following 7-weeks of intervention use.
  Assesses self-reported use and residual disability with 'old' hearing aids (Part I), as well as use and residual disability with 'new' hearing aids, and the difference in benefit and and satisfaction between 'old and 'new' hearing aids (Part II). Each domain is measured on a five-point scale.
Auditory Lifestyle and Demands Questionnaire | Following 1-week of intervention use.
  Self-report measure of auditory lifestyle.
Clarity and Comfort Questionnaire | Following 1-week of intervention use.
  Self-report measure of hearing aid preferences concerning sound clarity and comfort.
Hearing aid datalogging | Following 1-week and 7-weeks of intervention use.
  Hearing aid use in hours, internal to the hearing aid.
Montreal Cognitive Assessment | Following 1-week of intervention use.
  Validated screening tool for mild cognitive impairment.
BKB Speeh-In-Noise Test | Following 1-week and 7-weeks of intervention use.
  Behavioural measure of speech intelligibility in the presence of background noise.
eAdjust 0.2 app datalogging | Following 2-week and 6-weeks of intervention use.
  Usage data, internal to the app.
App real-world use questionnaire | Following 2-week and 6-weeks of intervention use.
  Self-report questionnaire of app usage. Consists of closed- and open-ended questions.
Hearing aid tasks | Following 2-week and 6-weeks of intervention use.
  Self-report questionnaire of app functionality in different environments.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute for Health Research Nottingham Biomedical Research Centre, Nottingham, Non-US/Non-Canadian, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gomez R, Habib A, Maidment DW, Ferguson MA. Smartphone-Connected Hearing Aids Enable and Empower Self-Management of Hearing Loss: A Qualitative Interview Study Underpinned by the Behavior Change Wheel. Ear Hear. 2022 May/Jun;43(3):921-932. doi: 10.1097/AUD.0000000000001143. PMID 34653030